CLINICAL TRIAL: NCT06665308
Title: Cognitive Status, Fatigue, and Inflammation in Patients With Immune Thrombocytopenic Purpura (ITP)
Brief Title: Cognitive Status, Fatigue and Inflammation in Patients With Immune Thrombocytopenia (ITP)
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18052; U1111-1299-2041 (Other: ICTRP)
Record Dates: First submitted 2024-10-10; First posted 2024-10-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Immune Thrombocytopenia; Primary Immune Thrombocytopenia; Adult Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention will be administered to study participants. Data will be collected using a combination of chart review, clinical outcome assessment administration, and laboratory results through blood tests.

SUMMARY:
This is a multi-center, hospital based, cross-sectional study based on data from patient medical records, including laboratory results. The study will include adult patients with chronic (> 1 year duration) primary Immune Thrombocytopenia (ITP) only. Patients will be identified based on a laboratory confirmed diagnosis of ITP in the medical records, where there is also a physician-confirmed diagnosis of primary ITP. If patients consent to take part in the study, a routine clinical visit will also serve as the study visit. Patients who do not have a routine visit scheduled during the study period but who would otherwise be eligible may be contacted by the site. In such cases, clinicians may use their discretion to schedule a visit specifically for study purposes.

All study participants will have a routine blood test as part of their standard clinical care at the study visit, and this same procedure will be used to collect supplementary blood samples to assess a variety of biomarkers.

Data will be collected using a combination of chart review, clinical outcome assessment administration, and laboratory results through blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with chronic (ITP with > 1 year duration) primary ITP living in the USA or the UK:

  * On ITP pharmacologic treatment, , including on-demand treatment strategy, regardless of last platelet count (below or above 100 x 10^9 counts/L);
  * Patients with their most recent platelet count >50 x 109 counts/L) and without any ITP-specific treatment for 1 year or less.
* Adult patient who are 18 years or older at index date
* Patient who has received at least one initial first line ITP therapy (CS/ IVIg/ANTI d) with initial response as of index date and indicated by one of the following:

  * Platelet count ≥ 50 x 10^9 counts /L; OR
  * Platelet count ≥ 30 x 10^9 counts /L with at least a two-fold increase from baseline within 1 month since start of treatment, as per ASH 2019 guidelines; OR
  * A medical record of initial response as determined by clinical judgement, considering documented platelet count along with overall patient condition and relevant medical factors.
* Patients whose medical history related to the study objectives are available from the site covering 12 months prior to index date.
* Patient provided informed consent to participate in the study.

Exclusion Criteria:

* Secondary ITP.
* Patients with their most recent platelet count >50 x 10^9 counts/L and without any ITP-specific treatment for more than 1 year.
* Patients with recent or active infection recorded 14 days or less before index date; patients with uncontrolled chronic infections or who were recently diagnosed with a chronic infection (≤14 days of index date).
* Patients with vaccination in 28 days before index date.
* Patients treated with rilzabrutinib on or before index date.
* Patients who participated in an interventional clinical trial for any investigational drug in the 180 days prior to index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this study will be patients treated for primary chronic Immune Thrombocytopenia at one of the four study centers in two countries (3 centers in the USA, 1 center in the UK).
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of impaired cognitive status among adult Immune Thrombocytopenia patients | Day 1 (Index date)
  Impaired cognitive status is defined as a CBB (CogState Brief Battery) z-score of -1 or less on at least one of 2 composite domains (attention/psychomotor composite and memory/learning composite domains).
  The CBB is a computerized outcome measure of cognitive function in human subjects aged 6 to 99 years and has been previously used in ITP. The CBB test for psychomotor function, attention, visual learning and working memory.

SECONDARY OUTCOMES:
Age, sex, ethnicity, educational attainment | Day 1 (Index date)
Smoking, alcohol, marijuana, cocaine use | Day 1 (Index date)
Comorbidities at index categorical | Day 1 (Index date)
Current medications | Day 1 (Index date)
  ITP-specific treatments, antiplatelet,anticoagulant, psychiatric and pain medications
ITP-PAQ | Day 1 (Index date)
  A validated, disease-specifictool to measure health-related quality of life HRQoL in adult ITP patients
ITP Bleeding Scale (IBLS) | Day 1 (Index date)
Medical history | Day 1 (Index date)
  Family history of dementia, family history of cognitive impairment, ITP medication and treatment history, age of ITP diagnosis, duration of ITP, history of clinically relevant or severe bleeding complications, history of thromboembolism complications, history of brain injury or neurological sequalae, history of COVID-19, brain imaging results, platelet counts results
Laboratory characteristics | Day 1 (Index date)
  Complete Blood Count
Assessment of key inflammatory biomarkers | Day 1 (Index date)
  Transferrin, Ferritin, Iron, Prothrombin fragment, Fibrinogen, D dimer, Interleukin (IL)-1 beta, IL-6, IL-10, IL-18, TNF alpha, Gamma Interferon, high-sensitivity C-reactive protein (hsCRP), MCP1, NETosis markers (cell-free deoxyribonucleic acid (DNA), neutrophil elastase (NE), myeloperoxidase (MPO)), antinuclear antibodies (ANA), Lupus anticoagulant, Anticardiolipin antibodies (ACA), thrombopoietin level, soluble P-selectin, L-selectin, ICAM-1; whole blood RNA sequencing (transcriptome), C1q, sC5b-9
FACIT (Functional Assessment of Chronic Illness Therapy) - Fatigue score | Day 1 (Index date)
  The FACIT-Fatigue is a 13-item tool that measures self-reported fatigue and its impact on daily life. Each question is rated by the participant on a Likert-like scale of 0 ('not at all') to 4 ('very much'). A higher FACIT-Fatigue score represents greater quality of life (QoL).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - USC Norris Comprehensive Cancer Center- Site Number : 8400002, Los Angeles, California
  - Massachusetts General Hospital- Site Number : 8400001, Boston, Massachusetts
  - University of Washington-Fred Hutchinson Cancer Center_Site Number: 8400003, Seattle, Washington
- Investigational Site Number: 8260001, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org